CLINICAL TRIAL: NCT02491099
Title: A Phase II Evaluation of Afatanib, an Irreversible Human Epidermal Growth Factor Receptor 2 (Her2/Neu) Tyrosine Kinase Inhibitor, in Patients With Persistent or Recurrent HER2-positive Uterine Serous Carcinoma
Brief Title: A Phase II Evaluation of Afatinib in Patients With Persistent or Recurrent HER2-positive Uterine Serous Carcinoma
Acronym: Afatinib
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1503015437
Record Dates: First submitted 2015-07-02; First posted 2015-07-07 (Estimated); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: HER2/Neu+ Uterine Serous Carcinoma
MeSH Terms: interventions — Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Afatinib (Experimental): Afatinib 40 mgs., Q 21 Day times 4 Cycles
  Interventions: Drug: Afatinib

INTERVENTIONS:
Drug: Afatinib — Afatinib, 40 mg orally once daily on a 21 day cycle for the first 12 weeks, then every 28 days for subsequent cycles until progression
  Other Names: Irreversible Human Epidermal Growth Factor

SUMMARY:
Primary Objective: To assess the activity of Afatinib in patients with persistent or recurrent uterine serous carcinoma overexpressing HER2/neu with the frequency of patients who survive progression-free for at least 6 months after initiating therapy. Secondary Objectives: To assess objective response rate and durable disease control rate. To assess overall survival. To assess the safety profile of Afatinib in uterine serous carcinoma patients.

DETAILED DESCRIPTION:
Exploratory/correlative objectives: To systematically evaluate HER2/neu expression/amplification using standardized scoring criteria for both breast and gastric cancer and correlate clinical response in uterine serous carcinoma patients with HER2/neu scoring results. To correlate objective response rate, PFS and overall survival with the presence/absence of phosphatidyl inositol 3-kinase catalytic subunit and F-box/WD repeat-containing protein mutations by standard Sanger sequencing, and presence/absence of Cyclin E2 overexpression by IHC in endometrial cancer patients overexpressing HER2/neu treated with Afatinib. To study HER2/neu extracellular domain circulating levels in the plasma of uterine serous carcinoma patients overexpressing HER2/neu before and during Afatinib treatment to elucidate whether changes in HER2/neu extracellular domain would predict response to Afatinib and to determine peripheral blood natural killer cell numbers and activity in HER2/neu+ uterine serous carcinoma patients before and during Afatinib treatment to assess the possible therapeutic contributions of immune mechanisms of action of Afatinib.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have persistent or recurrent histologically confirmed uterine serous carcinoma, harbor a tumor HER2/neu+ based upon IHC staining score of 3+ or 2+ with confirmed gene amplification by FISH.
* Have measurable disease.
* Have at least one target lesion to be used to assess response as defined by RECIST v1.1.
* After undergoing surgery may be optimally or sub optimally debulked, with measurable recurrent disease of any previous substage.
* Diagnosis histologically confirmed by a gynecologic pathologist as containing >10% uterine papillary serous adenocarcinoma in the specimen.
* Have adequate bone marrow function.
* WBC greater than or equal to 3,000/ul, platelets greater than or equal to 75,000/ul, neutrophils greater than or equal to 1500/ul., creatinine less than or equal to 2.0 mg/kl, bilirubin < 1.5 X laboratory normal, SGOT/SGPT <3 X laboratory normal.
* Have an ECOG performance status of 0 or 1.
* Have signed an approved consent.
* Have recovered from effects of recent surgery, radiotherapy or chemotherapy. Should be free of significant infection.
* Patients with recurrent disease may have received multiple prior chemotherapies for treatment of their uterine cancer.
* May have received prior trastuzumab therapy alone or in combination with chemotherapy with 2 week washout period required between trastuzumab treatment and first dose of Afatanib.
* Patients of childbearing potential must have a negative serum pregnancy test within 7 days prior to the study entry and be practicing an effective form of contraception.
* Must be 18 years of age.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial. NOTE: Patients with prior anthracycline exposure are NOT eligible.

Exclusion Criteria:

* Patients who have a significant history of cardiac disease, uncontrolled hypertension, unstable angina, uncontrolled congestive heart failure, or uncontrolled arrhythmias within 6 months of registration. Patients with any unstable medical issue, active treatment for symptomatic pulmonary embolism, CVA, renal or hepatic insufficiency, active infection/sepsis requiring IV antibiotics, known brain/leptomengial involvement of the disease, active neurological disease, dementia.
* Patients who have received prior therapy with any irreversible human epidermal growth factor receptor tyrosine kinase inhibitor.
* Patients who have an uncontrolled seizure disorder or active neurological disease. Patients known to be seropositive for HIV and active hepatitis, even if liver function studies are in the eligible range. Known hemorrhagic diathesis or active bleeding disorder.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-06; Primary Completion 2026-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 4 Years
  Progression free survival for at least 6 months after initiating therapy

SECONDARY OUTCOMES:
The safety profile of Afatinib in USPC patients by CTCAE v4.0 | 4 Years

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Santin, M.D., Principal Investigator — Yale University
Locations (3):
- United States (3):
  - University of Arizona Cancer Center, Tucson, Arizona
  - Yale New Haven Hospital, New Haven, Connecticut
  - Massachusetts General Hospital, Boston, Massachusetts

REFERENCES:
- [Result] Santin AD, Bellone S, Gokden M, Palmieri M, Dunn D, Agha J, Roman JJ, Hutchins L, Pecorelli S, O'Brien T, Cannon MJ, Parham GP. Overexpression of HER-2/neu in uterine serous papillary cancer. Clin Cancer Res. 2002 May;8(5):1271-9. PMID 12006548
- [Result] Santin AD, Bellone S, Van Stedum S, Bushen W, De Las Casas LE, Korourian S, Tian E, Roman JJ, Burnett A, Pecorelli S. Determination of HER2/neu status in uterine serous papillary carcinoma: Comparative analysis of immunohistochemistry and fluorescence in situ hybridization. Gynecol Oncol. 2005 Jul;98(1):24-30. doi: 10.1016/j.ygyno.2005.03.041. PMID 15894362
- [Result] Zhao S, Choi M, Overton JD, Bellone S, Roque DM, Cocco E, Guzzo F, English DP, Varughese J, Gasparrini S, Bortolomai I, Buza N, Hui P, Abu-Khalaf M, Ravaggi A, Bignotti E, Bandiera E, Romani C, Todeschini P, Tassi R, Zanotti L, Carrara L, Pecorelli S, Silasi DA, Ratner E, Azodi M, Schwartz PE, Rutherford TJ, Stiegler AL, Mane S, Boggon TJ, Schlessinger J, Lifton RP, Santin AD. Landscape of somatic single-nucleotide and copy-number mutations in uterine serous carcinoma. Proc Natl Acad Sci U S A. 2013 Feb 19;110(8):2916-21. doi: 10.1073/pnas.1222577110. Epub 2013 Jan 28. PMID 23359684
- [Result] Cancer Genome Atlas Research Network; Kandoth C, Schultz N, Cherniack AD, Akbani R, Liu Y, Shen H, Robertson AG, Pashtan I, Shen R, Benz CC, Yau C, Laird PW, Ding L, Zhang W, Mills GB, Kucherlapati R, Mardis ER, Levine DA. Integrated genomic characterization of endometrial carcinoma. Nature. 2013 May 2;497(7447):67-73. doi: 10.1038/nature12113. PMID 23636398
- [Result] Schwab CL, Bellone S, English DP, Roque DM, Lopez S, Cocco E, Nicoletti R, Bortolomai I, Bonazzoli E, Ratner E, Silasi DA, Azodi M, Schwartz PE, Rutherford TJ, Santin AD. Afatinib demonstrates remarkable activity against HER2-amplified uterine serous endometrial cancer in vitro and in vivo. Br J Cancer. 2014 Oct 28;111(9):1750-6. doi: 10.1038/bjc.2014.519. Epub 2014 Sep 30. PMID 25268372
- [Result] Santin AD, Bellone S, Siegel ER, Palmieri M, Thomas M, Cannon MJ, Kay HH, Roman JJ, Burnett A, Pecorelli S. Racial differences in the overexpression of epidermal growth factor type II receptor (HER2/neu): a major prognostic indicator in uterine serous papillary cancer. Am J Obstet Gynecol. 2005 Mar;192(3):813-8. doi: 10.1016/j.ajog.2004.10.605. PMID 15746676